CLINICAL TRIAL: NCT05757297
Title: Gut Microbiota and Failure of Endovascular Revascularization in Diabetic Patients With Peripheral Arterial Disease and Chronic Limb-threatening Ischemia
Brief Title: Gut Microbiota in Patients With Peripheral Arterial Disease and Chronic Limb-threatening Ischemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Flex Andrea, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5200
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Arterial Disease
Keywords: microbiota; gut microbiota; TMAO; MACE; MALE
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Microbiota has been associated with risk factors for cardiovascular diseases (hypertension, obesity, dyslipidemia, diabetes mellitus, heart failure). In animal models, the gut microbiota produces pro-inflammatory proteoglycans that increase the extent of myocardial infarction, reduced by treatment with probiotics (Lactobacillus). TMAO, a blood metabolite directly dependent on the gut microbiota is related to atherosclerotic plaque instability and major adverse cardiovascular events (MACE) in humans. Recent data demonstrate that blood levels of TMAO directly correlate with the risk of major MACE and mortality in patients with peripheral arterial disease (PAD).

The goal of this observational study is to evaluate the association between gut microbiota and TMAO serum levels and MACE and major adverse limb events (MALE) in patients with PAD and chronic limb threatening ischemia (CLTI) requiring a procedure of endovascular revascularization.

The main questions it aims to answer are:

* association between gut microbiota and TMAO serum levels and MALE after lower extremity revascularization.
* association between gut microbiota and TMAO serum levels and MACE after lower extremity revascularization.

Patients with CLTI requiring lower extremity endovascular revascularization will undergo stool sampling for determination of gut microbiota and blood sampling for the dosage of circulating TMAO before the endovascular procedure.

Incidence of MALE and MACE will be collected in a 24-months follow-up and will be associated with gut microbiota and TMAO serum levels.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 18 years
* Ankle/Brachial Index (ABI) of less than 80
* at least one lower limb stenosis greater than 50% documented by Ultrasound Color Doppler (US)
* stage 4 or 5 PAD diagnosis according to the Rutherford classification
* presence of chronic limb-threatening ischemia
* indication for LER of the target arterial stenosis

Exclusion Criteria:

* acute infections at present or in the previous month
* antibiotic treatment in the previous month
* primary hyperparathyroidism
* revascularization of the lower limb in the previous 3 months
* diabetic foot ulcers with signs of active infection or osteomyelitis
* organ transplantation
* active cancer
* liver disease at functional status B or C according to Child-Pugh
* absolute contraindication to antiplatelet therapy
* thrombophilia
* contraindication to endovascular revascularization

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will enroll consecutive subjects with PAD and CLTI requiring for endovascular revascularization and admitted to Internal Medicine Cardiovascular Unit of the Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Association between incidence of MALE and gut microbiota and TMAO serum levels | 24-months follow-up
  To evaluate the association between gut microbiota and TMAO serum levels before endovascular revascularization and incidence of MALE during the follow-up period.

SECONDARY OUTCOMES:
Association between incidence of myocardial infarction and gut microbiota and TMAO serum levels | 24-months follow-up
  To evaluate the association between gut microbiota and TMAO serum levels before endovascular revascularization and incidence of myocardial infarction during the follow-up period.
Association between incidence of stroke and gut microbiota and TMAO serum levels | 24-months follow-up
  To evaluate the association between gut microbiota and TMAO serum levels before endovascular revascularization and incidence of stroke during the follow-up period.
Association between incidence of cardiovascular death and gut microbiota and TMAO serum levels | 24-months follow-up
  To evaluate the association between gut microbiota and TMAO serum levels before endovascular revascularization and incidence of cardiovascular death during the follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy